CLINICAL TRIAL: NCT00702416
Title: Ultrasound Guidance or Electrical Nerve Stimulation for Interscalene Brachial Plexus Block: a Randomized, Controlled Trial
Brief Title: Ultrasound Guidance for Interscalene Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Guido Fanelli, MD, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANEST-ORT-01
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Shoulder; Orthopedic Surgery; Nerve Block
Keywords: Analgesia, Patient-controlled; Anesthesia, Regional; Ultrasound; Postoperative Pain; Brachial Plexus
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — High-Energy Shock Waves; Anesthesia, Conduction; Transcutaneous Electric Nerve Stimulation; Ropivacaine; Anesthetics, Local; Acetaminophen; Analgesics; Morphine; Analgesics, Opioid; Narcotics; Fentanyl; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- US Group (Experimental): In this group, the continuous block will be performed under real-time ultrasound (US) guidance.
  Interventions: Procedure: Ultrasound-guided continuous interscalene brachial plexus block; Drug: Ropivacaine; Drug: Paracetamol; Drug: Morphine; Drug: Fentanyl; Procedure: General anesthesia
- ENS Group (Active Comparator): In this group, the continuous block will be performed with an electrical nerve stimulation (ENS) technique.
  Interventions: Procedure: Continuous interscalene brachial plexus block using electrical nerve stimulation; Drug: Ropivacaine; Drug: Paracetamol; Drug: Morphine; Drug: Fentanyl; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Ultrasound-guided continuous interscalene brachial plexus block — With patients in the supine position, a high-frequency (10-12 MHz) ultrasound transducer in a sterile sheath will be applied to explore the interscalene region and locate the brachial plexus. The transducer will be positioned so as to image the C5 and C6 roots in a single view. Visualization of the C7 root in the same scan will be sought, but will not be required.
  A 50-mm, 20 G needle will be advanced in-plane from the postero-lateral side of the transducer. Injection of the local anesthetic will be performed in small aliquots while repositioning of the needle in order to optimize spread of the injectate around the nerve roots.
  At the end of the injection, a catheter will be threaded through the needle. The catheter will be positioned to lie deep and close to the imaged nerve roots.
  Other Names: Peripheral nerve block; Ultrasound; Regional anesthesia
  Arms: US Group
Procedure: Continuous interscalene brachial plexus block using electrical nerve stimulation — With patients in the supine position, the head will be rotated to the contralateral side. The interscalene groove will be palpated.
  A 35-mm, 20 G needle will be inserted at the estimated C6 level (cricoid cartilage) with a 30-45° angle to the skin. The needle will be advanced along a line joining the insertion site to the axilla.
  An electrical nerve stimulator will be used at an initial intensity of 1.0 mA (frequency: 2 Hz, pulse width: 0.2 ms). A musculocutaneous or axillary-nerve mediated twitch will be sought
  Injection of the local anesthetic will start with a visible motor response at a current <0.5 mA. The catheter will be positioned to as to elicit a motor response at ≤0.4 mA.
  Other Names: Peripheral nerve block; Electrical nerve stimulation; Regional anesthesia
  Arms: ENS Group
Drug: Ropivacaine — Block induction [1% (wt/vol) solution]:
  20 ml (200 mg)
  Postoperative analgesia [0.2% (wt/vol) solution]:
  * Background infusion: 4 ml/h (8 mg/h)
  * Incremental on-demand dose: 2 ml (4 mg)
  * Lockout time: 15 min
  Other Names: Naropin; Local anesthetic; Amide local anesthetic
Drug: Paracetamol — 1 g iv q8h
  Other Names: Acetaminophen; Perfalgan; Analgesic
Drug: Morphine — 5 mg im prn q1h (in the postoperative period)
  Other Names: Opioid; Narcotic; Analgesic
Drug: Fentanyl — 50 µg iv prn (in the intraoperative period)
  Other Names: Opioid; Narcotic; Analgesic
Procedure: General anesthesia — Will be given in case of block failure and/or patient discomfort intractable with fentanyl during the procedure.
  The technique will be left at the discretion of the attending anesthesiologist. Monitored anesthesia care will also be acceptable; the block will be considered as failed in that case as well.
  Other Names: Monitored anesthesia care

SUMMARY:
This study has been designed to assess the possible advantages of using ultrasound imaging to block the brachial plexus (i.e., nerves of the upper limb) in patients undergoing shoulder surgery.

The ultrasound technique will be compared with the current gold standard, electrical nerve stimulation.

The aim of this study is to define which technique is better in terms of time to onset of anesthesia.

DETAILED DESCRIPTION:
The study will compare real-time ultrasound (US) guidance and electrical nerve stimulation (ENS) in terms of onset time for interscalene brachial plexus anesthesia.

The main hypothesis is that direct visualization of neural structures under US guidance will grant better local anesthetic (LA) disposition around the roots of the plexus, thus improving onset times.

Perineural catheters will be used to maintain regional analgesia for 48 hours after surgery. We hypothesize that US guidance may also help physicians place perineural catheters more precisely, thus improving analgesia in the following hours to days.

Finally, we will investigate for possible differences in minor adverse events such as vascular puncture, pain during the anesthetic procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status Class I-III
* Elective surgery of the shoulder
* Informed consent to regional anesthesia

Exclusion Criteria:

* Inability to effectively communicate
* Chronic opioid use
* Absence of informed consent to participation to the study
* Ipsilateral upper limb neurological deficits
* Known allergy to study medications
* Contraindications to continuous block placement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Onset time of brachial plexus anesthesia | ≤30 min

SECONDARY OUTCOMES:
Successful brachial plexus anesthesia | ≤30 min
Additional analgesic requirements during surgery | Duration of surgery
Incidence of paresthesiae during the anesthetic procedure | ≤30 min
Incidence of blood aspiration during the anesthetic procedure | ≤30 min
Number of needle redirections for the performance of the block | ≤30 min
Pain during performance of the block | ≤30 min
Pain at rest and on movement (visual analog scale) | q8h until 48 h after surgery
Local anesthetic consumption on patient-controlled pump | ≤48 h

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Danelli, MD, Principal Investigator — UO II Anestesia, Rianimazione e Terapia Antalgica, AOU Parma
Locations (1):
- University Hospital / Azienda Ospedaliero-Universitaria, Parma, PR, Italy

REFERENCES:
- [Background] Casati A, Fanelli G, Aldegheri G, Berti M, Colnaghi E, Cedrati V, Torri G. Interscalene brachial plexus anaesthesia with 0.5%, 0.75% or 1% ropivacaine: a double-blind comparison with 2% mepivacaine. Br J Anaesth. 1999 Dec;83(6):872-5. doi: 10.1093/bja/83.6.872. PMID 10700785
- [Background] Stevens MF, Werdehausen R, Golla E, Braun S, Hermanns H, Ilg A, Willers R, Lipfert P. Does interscalene catheter placement with stimulating catheters improve postoperative pain or functional outcome after shoulder surgery? A prospective, randomized and double-blinded trial. Anesth Analg. 2007 Feb;104(2):442-7. doi: 10.1213/01.ane.0000253513.15336.25. PMID 17242107
- [Background] Casati A, Borghi B, Fanelli G, Montone N, Rotini R, Fraschini G, Vinciguerra F, Torri G, Chelly J. Interscalene brachial plexus anesthesia and analgesia for open shoulder surgery: a randomized, double-blinded comparison between levobupivacaine and ropivacaine. Anesth Analg. 2003 Jan;96(1):253-9, table of contents. doi: 10.1097/00000539-200301000-00051. PMID 12505962
- [Background] Casati A, Danelli G, Baciarello M, Corradi M, Leone S, Di Cianni S, Fanelli G. A prospective, randomized comparison between ultrasound and nerve stimulation guidance for multiple injection axillary brachial plexus block. Anesthesiology. 2007 May;106(5):992-6. doi: 10.1097/01.anes.0000265159.55179.e1. PMID 17457131